CLINICAL TRIAL: NCT06234696
Title: The Effect of Based Cognitive Behavioral Therapy by Humor Based Psychoeducation on Sense of Humour, Self Esteem and Depression Levels Patient in Diagnosed With Depression
Brief Title: Cognitive Behavioral Therapy by Humor Based Psychoeducation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Fatima Ozdemir Sigva, Psychiatric Nurse, University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AIBU-SBF-FŞ-1
Record Dates: First submitted 2024-01-04; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Depression
Keywords: cognitive behavioral therapy; depression; humor
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The group consists of 30 people and this group will be given psychoeducation for 4 weeks.
  Training will be provided 2 days a week (monday and friday).
  Interventions: Other: entrepreneurial intervention
- control group (No Intervention): The group consists of 30 people and this group will not be trained.

INTERVENTIONS:
Other: entrepreneurial intervention — The experimental group will be given psychoeducation for 4 weeks.
  Arms: experimental group

SUMMARY:
This study aims to reveal the effectiveness of based cognitive behavioral therapy by humor based psychoeducation on sense of humour, self-esteem and depressıon level patient in diagnosed with deppression .

DETAILED DESCRIPTION:
Aim: This study aims to reveal the effectiveness of based cognitive behavioral therapy by humor based psychoeducation on sense of humour, self esteem and depression level patient in diagnosed with depression .

Method: This study will be conducted as a randomized controlled experimental study by the researcher, who is a specialist psychiatric nurse, to the elderly patient in diagnosed with depression staying in the mardin traning and research hospital and kızıltepe state hospital. In the study, "power analysis" was performed and a total of 44 individuals, including 22 intervention people and 22 control group, were considered suitable for the sample size. It was decided to have 30 people in the groups, considering the high power of the test and the loses in the study. Accordingly, 30 people were determined as the intervention group and 30 people as the control group. In this study, personal ınformation form, coping humor scale, rosenberg self-esteem scale, beck depression scale, multidimensional sense of humor scale.

Findings: Aims to reveal the effectiveness of based cognitive behavioral therapy by humor based psychoeducation on sense of humour, self esteem and depression levels patient in diagnosed with depression .

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Not having any obstacle to communication
* Being between the ages of 18 and 65
* Being monitored on an outpatient basis with a diagnosis of depression according to the diagnostic and statistical manual of mental disorders criteria
* Being literate
* Not having undergone such training in the last 6 months

Exclusion Criteria:

* Serious factors that may prevent you from answering the survey
* Presence of physical and cognitive disability
* Refusing to participate in the study after being informed
* Having a comorbid psychiatric diagnosis
* A patient diagnosed with depression with psychotic features
* Having received any psychotherapy in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-30 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Data Collection Tools Personel İnformation Form | Between 1-3 months
  Data Collection Tools Personel İnformation Form: form, organised by the researchers, includes 16 questions to determine the demograhic information of the participants.
Coping humor scale | Between 1-3 months
  Coping humor scale: The scale is a 4-point Likert-tybe scale (1: Strongly disagree - 4: Completely agree) consisting of 7 items. The lowest score to be obtained from the scale 7 and the highest score is 28. Rising scores indicate that individuals have a higher level of ability to use humor as a coping strategy in stressful situations.
Multidimensional sense of humor scale | Between 1-3 months
  Multidimensional sense of humor scale:The scale consists of a total of 24 items and four subscales. The items in the scale are avaluated using 5- point likert tybe scale (0= strongly disagree, 4 = strongly agree) The lowest score to be obtained from the scale 0 and the highest score is 96.In addition to a general sense of humor score, the scale has 4 subscales: producing humor, coping using humor, attitude towards people who produce humor, and humor evaluation.
Rosenberg self-esteem scale | Between 1-3 months
  Rosenberg self-esteem scale: The scale consists of total 63 items and 12 subscales.In our study, only the part of the scale related to self-esteem will be used. The self-esteem subscale is a Likert-type subscale consisting of 4 items and includes the first 10 items of the inventory. Each statement contains 4-point Likert type options (4=very true, 3=true,2= false,1= very false). When evaluating, in positive statements, the "very true" option is 4 points, the "very wrong" option is 1 point; For negative expressions, the calculation was made exactly the opposite. Depending on the evaluation method of the scale, 0-6 points can be obtained. Thus, the person who completes the test can get a maximum of 6 points in total. 5-6 points were determined as low self-esteem, 2-4 points as medium self-esteem, and 0-1 points as high self-esteem.
Beck depression scale | Between 1-3 months
  Beck depression scale: This scale consists of 21 items and each item has four options. The four options in each symptom category of the scale receive a score between 0 and 3. The highest score that can be obtained from the scale is 63. A high total score indicates a high level or severity of depression symptoms.10-17 points from the scale indicate mild depression, 18-29 points indicate moderate depression, and 30-63 points indicate severe depression.
Data Analysis | Between 1-3 months
  Data Analysis: The data obtained from the study will be analysed in Statistical Packkage for Social Sciences 22 package programme. Repeated Measures Analysis Of Variance was used to compare the scale scores and Fisher Least Significant Difference test was used for multiple comparisons of Group Time interaction

CONTACTS AND LOCATIONS:
Overall Officials: nurgül özdemir, Study Director — 05332352154
Locations (1):
- Fatima, Mardin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes